CLINICAL TRIAL: NCT02619994
Title: Delamanid, Linezolid, Levofloxacin, and Pyrazinamide for the Treatment of Patients With Fluoroquinolone-sensitive MDR-TB: A Phase 2/3, Multicenter, Randomized, Open-label, Clinical Trial
Brief Title: Treatment Shortening of MDR-TB Using Existing and New Drugs
Acronym: MDR-END
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Dankook University (Other); International Tuberculosis Research Center (Other); Pusan National University Yangsan Hospital (Other); Pusan National University Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); SMG-SNU Boramae Medical Center (Other); Incheon St.Mary's Hospital (Other); Ulsan University Hospital (Other); Korean Institute of Tuberculosis (Other); National Medical Center, Seoul (Other); Korean Center for Disease Control and Prevention (Other Government); Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDR-END
Record Dates: First submitted 2015-11-24; First posted 2015-12-02 (Estimated); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: Multidrug-resistant tuberculosis; Linezolid; Delamanid; Multicenter randomized trial; Non-inferiority; Shorter regimen
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Linezolid; OPC-67683; Levofloxacin; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Active Comparator): Regimen is the locally-used WHO-approved MDR-TB regimen in Korea based on 2014 Korean guideline of TB management.
  * Intensive phase regimen consists of four effective second-line anti-TB drugs (including injectables) and pyrazinamide.
  * Treatment duration: for at least 20 months
  Interventions: Drug: Locally-used WHO-approved MDR-TB regimen in Korea
- Experimental Arm (Experimental): Regimen consists of only oral medication using delamanid, linezolid, levofloxacin, and pyrazinamide, for nine or twelve months depending on the time of sputum culture conversion to negative.
  * Delamanid (100 mg bid for the entire treatment period)
  * Linezolid (600mg/day for 2 months and 300mg/day afterwards until the end of treatment)
  * Levofloxacin (750 ~1000 mg/day)
  * Pyrazinamide (1000~ 2000 mg/day)
  Interventions: Drug: Linezolid; Drug: Delamanid; Drug: Levofloxacin; Drug: Pyrazinamide

INTERVENTIONS:
Drug: Linezolid
  Arms: Experimental Arm
Drug: Delamanid
  Arms: Experimental Arm
Drug: Levofloxacin
  Arms: Experimental Arm
Drug: Pyrazinamide
  Arms: Experimental Arm
Drug: Locally-used WHO-approved MDR-TB regimen in Korea
  Arms: Control Arm

SUMMARY:
The purpose of this study is to compare the efficacy of a 'new treatment regimen including delamanid, linezolid, levofloxacin, and pyrazinamide for nine or twelve months (investigational arm)' and 'the standard treatment regimen including injectables for 20 to 24 months (control arm)' for treating fluoroquinolone-sensitive multidrug-resistant tuberculosis.

DETAILED DESCRIPTION:
This study is a phase II/III, multicenter, randomized, open-label clinical trial of non-inferiority design comparing a new regimen to the World Health Organization-endorsed conventional regimen for fluoroquinolone-sensitive MDR-TB. The control arm uses a conventional treatment regimen with second-line drugs including injectables for 20-24 months. The investigational arm uses a new shorter regimen including delamanid, linezolid, levofloxacin, and pyrazinamide for 9 or 12 months depending on time to sputum culture conversion. The primary outcome is the treatment success rate at 24 months after treatment initiation. Secondary outcomes include time to sputum culture conversion on liquid and solid media, proportions of sputum culture conversion on liquid media after 2 and 6 months of treatment, treatment success rate according to pyrazinamide resistance, and occurrence of adverse events grade 3 and above as evaluated by the Common Terminology Criteria for Adverse Events. The population number is calculated as 102 per group (204 in total).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged from 19 to 85 years
* Confirmed MDR-TB or RR-TB
* On current TB therapy for ≤14 days at the time of enrollment.

Exclusion Criteria:

* Known any quinolone-resistant MDR-TB
* Known XDR-TB
* who are pregnant or who are unwilling to use proper contraceptives at childbearing age
* Medical history of galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* The need for ongoing use of prohibited drugs while on study drugs
* History of optic neuropathy or peripheral neuropathy
* With any of the following test results: i.Absolute neutrophil count < 2000 cells/mL, ii.White blood cell count (WBC) < 3.0 X 103/µL, iii.Hemoglobin < 7.0 g/dL, iv.Serum creatinine > 2.0 mg/dL, v.Aspartate aminotransferase (AST or SGOT) >100 IU/L, vi.Alanine aminotransferase (ALT or SGPT) >100 IU/L, vii.Total bilirubin > 2.0 mg/dL, viii.Albumin < 2.8g/dL, ix.QTcF > 500ms
* History of hypersensitivity reaction to the study drugs

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Mok J, Lee M, Kim DK, Kim JS, Jhun BW, Jo KW, Jeon D, Lee T, Lee JY, Park JS, Lee SH, Kang YA, Lee JK, Kwak N, Ahn JH, Shim TS, Kim SY, Kim S, Kim K, Seok KH, Yoon S, Kim YR, Kim J, Yim D, Hahn S, Cho SN, Yim JJ; MDR-END investigators. 9 months of delamanid, linezolid, levofloxacin, and pyrazinamide versus conventional therapy for treatment of fluoroquinolone-sensitive multidrug-resistant tuberculosis (MDR-END): a multicentre, randomised, open-label phase 2/3 non-inferiority trial in South Korea. Lancet. 2022 Oct 29;400(10362):1522-1530. doi: 10.1016/S0140-6736(22)01883-9. PMID 36522208
- [Derived] Lee M, Mok J, Kim DK, Shim TS, Koh WJ, Jeon D, Lee T, Lee SH, Kim JS, Park JS, Lee JY, Kim SY, Lee JH, Jo KW, Jhun BW, Kang YA, Ahn JH, Kim CK, Shin S, Song T, Shin SJ, Kim YR, Ahn H, Hahn S, Won HJ, Jang JY, Cho SN, Yim JJ. Delamanid, linezolid, levofloxacin, and pyrazinamide for the treatment of patients with fluoroquinolone-sensitive multidrug-resistant tuberculosis (Treatment Shortening of MDR-TB Using Existing and New Drugs, MDR-END): study protocol for a phase II/III, multicenter, randomized, open-label clinical trial. Trials. 2019 Jan 16;20(1):57. doi: 10.1186/s13063-018-3053-1. PMID 30651149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 443 eligible patients, 229 were excluded for the following reasons:
  * By the investigators' decision (n=102)
  * Declined to participate (n=65)
  * Met one of the exclusion criteria (n=58)
  * Laboratory abnormalities (n=42)
  * Ongoing use of prohibited drugs (n=10)
  * Unwilling to use proper contraceptives (n=3)
  * History of optic or peripheral neuropathy (n=3)
  * Other unspecified reason (n=4)
Groups:
- Control Arm: Regimen is the locally-used WHO-approved MDR-TB regimen in Korea based on 2014 Korean guideline of TB management.
  * Intensive phase regimen consists of four effective second-line anti-TB drugs (including injectables) and pyrazinamide.
  * Treatment duration: for at least 20 months
  Locally-used WHO-approved MDR-TB regimen in Korea
- Experimental Arm: Regimen consists of only oral medication using delamanid, linezolid, levofloxacin, and pyrazinamide, for nine or twelve months depending on the time of sputum culture conversion to negative.
  * Delamanid (100 mg bid for the entire treatment period)
  * Linezolid (600mg/day for 2 months and 300mg/day afterwards until the end of treatment)
  * Levofloxacin (750 ~1000 mg/day)
  * Pyrazinamide (1000~ 2000 mg/day)
  Linezolid
  Delamanid
  Levofloxacin
  Pyrazinamide
Period: Overall Study
Arm/Group | Control Arm | Experimental Arm
Started | 106 | 108
Completed | 89 (mITT population) | 79 (mITT population)
Not Completed | 17 | 29

BASELINE CHARACTERISTICS:
Population: mITT population of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Experimental Arm | Total
Number analyzed (Participants) | 89 | 79 | 168
Age, Continuous [Median (Full Range); unit: years] | 46 [19 to 82] | 49 [19 to 85] | 47 [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 63 | 53 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 89 | 79 | 168
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 89 | 79 | 168
Baseline Characteristics of Participants [Count of Participants; unit: Participants] | 89 | 79 | 168

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Rate
Description: To test for non-inferiority of the investigational arm, when the lower limit of the one-sided 97.5% confidence interval of the difference (PT - PC) between investigational and control arms is larger than the non-inferiority margin of - 10%, it will be concluded that the treatment success rate of the investigational arm shows non-inferiority to the treatment success rate of the control arm.
  (primary consideration for the modified intention-to-treat results)
Time Frame: 24 months after treatment start
Population: mITT population Participant with [not assessable] was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 85 | 72
Participants | 60 | 54

2. Secondary Outcome: Time to Sputum Culture Conversion After Treatment Start
Description: To determine whether time to sputum culture conversion after treatment start is statistically different between the control and investigational arms, the median time will be estimated in each group using the Kaplan-Meier method, and the difference in the distribution of time to culture conversion of the two arms will be compared using the log-rank test.
Time Frame: through study completion (24 months after treatment start)
Population: Participants with a positive baseline M.tuberculosis culture (liquid media) in the mITT population
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 52 | 49
day | 24 [7 to 56] | 27 [7 to 55]

3. Secondary Outcome: Sputum Culture Conversion Proportion
Description: Culture conversion rate at month 2 of treatment in participants with positive baseline sputum culture (liquid media).
Time Frame: At 2 months of treatment
Population: mITT population Participants with positive baseline sputum culture
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 52 | 49
Participants | 42 | 35

4. Secondary Outcome: Treatment Success at the End of Treatment
Description: Treatment success rate at the end of treatment.
  * control arm (20-24 months)
  * experimental arm (40 or 52 weeks)
Time Frame: At the end of treatment
Population: mITT populration One participant of experimental arm who became pregnant during the treatment was excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 89 | 78
Participants | 64 | 61

5. Secondary Outcome: Proportion of Reverting to Positive Sputum Culture After the End of Treatment
Description: The proportion of patients who experienced a reversion between the end of treatment and up to 24 months after treatment start
Time Frame: At 24months after treatment start
Population: mITT population Participant with [not assessable] was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 85 | 72
Participants | 0 | 1

6. Secondary Outcome: Treatment Success According to Pyrazinamide Resistance (1)
Description: Treatment success rate of participants with pyrazinamide resistance in the mITT analysis
Time Frame: At 24months after treatment start
Population: mITT population Participant with [not assessable] was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 21 | 25
Participants | 13 | 19

7. Secondary Outcome: Proportion of Death Between the Control and Investigational Arms
Description: The proportion of participants who died in the control and experimental arm mITT population
Time Frame: At 24months after treatment start
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 89 | 79
Participants | 2 | 5

8. Secondary Outcome: Sputum Culture Conversion Proportion
Description: Culture conversion rate at month 6 of treatment in participants with positive baseline sputum culture (liquid media).
Time Frame: At 6 months of treatment start
Population: mITT population participants with positive baseline sputum culture (liquid media)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 52 | 49
Participants | 45 | 39

9. Secondary Outcome: Treatment Success According to Pyrazinamide Resistance (2)
Description: Treatment success rate of participants without pyrazinamide resistance in the mITT analysis
Time Frame: At 24 months after treatment start
Population: mITT population Participant with [not assessable] was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 52 | 42
Participants | 41 | 32

ADVERSE EVENTS:
Time Frame: All adverse events and serious adverse events were collected during the entire 24-month study period.
Description: Adverse Events were summarised according to the Common Terminology Criteria for Adverse Events
Arm/Group | Control Arm | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 2/89 | 5/79
Serious Adverse Events (participants affected / at risk) | 19/89 | 20/79
Other Adverse Events (participants affected / at risk) | 87/89 | 78/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=89) | Experimental Arm (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Cytopenia (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 4 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Computerised tomogram abnormal (Investigations) | 0 | 2
Hepatitis B DNA increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ligament operation (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=89) | Experimental Arm (N=79)
Anaemia (Blood and lymphatic system disorders) | 6 | 29
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 7 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 1
Diplopia (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Glare (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 1
Optic neuropathy (Eye disorders) | 0 | 3
Vision blurred (Eye disorders) | 8 | 5
Visual acuity reduced (Eye disorders) | 1 | 3
Visual impairment (Eye disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 5
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 15 | 19
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 25 | 16
Dysphagia (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 2 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Glossodynia (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 67 | 57
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 20 | 31
Asthenia (General disorders) | 4 | 7
Chest discomfort (General disorders) | 3 | 1
Chest pain (General disorders) | 5 | 0
Condition aggravated (General disorders) | 2 | 1
Fatigue (General disorders) | 5 | 3
Feeling hot (General disorders) | 2 | 1
Generalised oedema (General disorders) | 0 | 1
Granuloma (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 4
Pain (General disorders) | 3 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 4
Vessel puncture site bruise (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 9 | 2
Liver disorder (Hepatobiliary disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Dermatophytosis of nail (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 12 | 2
Otitis media (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Rash pustular (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 2 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 8 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 1
Blood bilirubin increased (Investigations) | 4 | 3
Blood creatinine increased (Investigations) | 2 | 7
Blood uric acid increased (Investigations) | 0 | 3
Colour vision tests abnormal (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 10
Hepatic enzyme abnormal (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 12 | 9
Neutrophil count decreased (Investigations) | 4 | 3
Platelet count decreased (Investigations) | 3 | 2
Weight decreased (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 12 | 15
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 5 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 21 | 20
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 11
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 18 | 8
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 9 | 21
Hypoaesthesia (Nervous system disorders) | 7 | 5
Lethargy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 15
Paraesthesia (Nervous system disorders) | 6 | 28
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Polyneuropathy (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 2 | 1
Delusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 5 | 5
Hallucination, visual (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 10 | 11
Major depression (Psychiatric disorders) | 1 | 0
Obsessive thoughts (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 19
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT02619994/Prot_SAP_000.pdf